CLINICAL TRIAL: NCT06359067
Title: A Real-World Study of Bispecific Antibodies, Teclistamab and Elranatamab, for Patients With Multiple Myeloma
Brief Title: A Real-World Study of Bispecific Antibodies in Multiple Myeloma
Acronym: BISPEMM
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240295
Record Dates: First submitted 2024-03-25; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Teclistamab; Elranatamab; Bispecific antibody
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treated by bispecific antibodies: Patients with multiple myeloma, penta-drug or triple class refractory and treated by bispecific antibodies, teclistamab or elranatamab
  Interventions: Other: Treated by bispecific antibodies, teclistamab or elranatamab in usual care
- Control group: Patients with multiple myeloma, penta-drug or triple class refractory and not treated by bispecific antibodies
  Interventions: Other: Not treated by bispecific antibodies in usual care

INTERVENTIONS:
Other: Treated by bispecific antibodies, teclistamab or elranatamab in usual care — Treated by bispecific antibodies, teclistamab or elranatamab in usual care
  Groups: Treated by bispecific antibodies
Other: Not treated by bispecific antibodies in usual care — Not treated by bispecific antibodies in usual care
  Groups: Control group

SUMMARY:
Bispecific antibody (BsAb) treatments, teclistamab and elranatamab, are newly available for patients with multiple myeloma who are refractory to all current drugs. The results are very encouraging but complicated adverse events, particularly infectious. This study analyzes survival data in patients treated with BsAb, as well as safety data, in particular the proportions and locations of infectious events. The results are compared to a control cohort. This study is multicentric on all the university hospitals of Paris (AP-HP).

DETAILED DESCRIPTION:
Bispecific antibody (BsAb) treatments, teclistamab and elranatamab, are newly available for patients with multiple myeloma who are refractory to all current drugs. The results are very encouraging but complicated adverse events, particularly infectious. This study analyzes survival data in patients treated with BsAb, as well as safety data, in particular the proportions and locations of infectious events. The results are compared to a control cohort. This study is multicentric on all the university hospitals of Paris (AP-HP).

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years old
* Patients with multiple myeloma
* Patients who received at least one administration of the following therapies: teclistamab, elranatamab

Exclusion Criteria:

- Patients opposed to the collection of their personal data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with multiple myeloma treated with bispecific antibodies, teclistamab or elranatamab.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Infection rate | Up to 18 months
  Explore the infection rate

SECONDARY OUTCOMES:
Global survival | Up to 18 months
  Explore the global survival
Progression-free survivals | Up to 18 months
  Explore the progression-free survivals

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie ZERBIT, PharmD, Principal Investigator — Pharmacy Department, Assistance Publique-Hopitaux de Paris, Université de Paris, Paris, France
Locations (1):
- Assistance Publique - Hôpitaux de Paris (AP-HP), Paris, IDF, France

IPD SHARING:
Plan to Share IPD: No